CLINICAL TRIAL: NCT04387851
Title: Learning Mechanisms for Placebo and Nocebo Studies on Somatosensory Sensations: a Systematic Review and Meta-analysis.
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Universiteit Leiden (Other)
Responsible Party: Principal Investigator, AWMEvers, Principal Investigator, Leiden University Medical Center
Other Study IDs: META-BLOM-DD-2022
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Pain; Itch
Keywords: Placebo; Nocebo; Pain; Itch; Somatosensory; Learning
MeSH Terms: conditions — Pain; Pruritus | interventions — Nocebo Effect

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Placebo: Placebo effects are defined as the positive effects occurring after the (supposed) administration of an inert treatment, which, through a given learning process, is believed to have positive effects.
  Interventions: Behavioral: Placebo induction; Behavioral: Control
- Nocebo: Nocebo effects are defined as the negative effects occurring after the (supposed) administration of an inert treatment, which, through a given learning process, is believed to have negative effects.
  Interventions: Behavioral: Control; Behavioral: Nocebo

INTERVENTIONS:
Behavioral: Placebo induction — The placebo interventions of interest are experimental learning methods (e.g. verbal suggestion, conditioning), used to induce placebo effects on somatosensory sensations.
  Groups: Placebo
Behavioral: Control — Placebo and nocebo effects should be measured relative to a control group (between-subjects design). In the case of within-subjects designs, these will be included to the extent possible (in a separate analysis or descriptively depending on the number of results).
Behavioral: Nocebo — The nocebo interventions of interest are experimental learning methods (e.g. verbal suggestion, conditioning), used to induce nocebo effects on somatosensory sensations.
  Groups: Nocebo

SUMMARY:
Placebo and nocebo effects are defined as the positive and negative effects occurring after the (supposed) administration of an inert treatment, which, through a given learning process, is believed to have positive or negative effects. The objective of this study is to summarize the available knowledge on experimental inductions of placebo and nocebo effects on somatosensory sensations, specifically pain and itch. The aim isto investigate the extent to which learning processes (such as conditioning and verbal suggestions) induce placebo and nocebo effects on pain and itch in healthy humans. The researchers intent to examine expectancy induction methods for placebo and nocebo effects on somatosensory sensations, describe methodological attributes of the research and propose practical and theoretical implications as well as future directions for research investigating placebo and nocebo effects on somatosensory sensations.

DETAILED DESCRIPTION:
Research questions include:

1. What is the average magnitude of placebo or nocebo effects on pain and on itch, across included studies?
2. Across studies that tested multiple learning processes for placebo and nocebo effects on pain, is the magnitude of a placebo or nocebo effect on pain different based on the learning process used to induce the effect?
3. Does the magnitude of placebo or nocebo effects differ between the sensations of pain and itch?
4. Are nocebo effects on pain and itch stronger than placebo effects on pain and itch, as measured by their relative magnitude?

Dependent upon search results, the researchers intend to answer questions 1 and 2 with meta-analysis, and questions 3 and 4 with systematic review.

Search Strategy:

PubMed, PsycINFO, EMBASE, and the Cochrane CENTRAL Methodology Library will be searched. Languages are restricted to English, Dutch, and German. Publication period is not restricted. Searches were initially conducted on March 18th, 2019. The detailed key-worded search strategy will not be made publicly available until this review is complete.

Condition or domain being studied:

Experimental induction of placebo or nocebo effects on somatosensory sensations (i.e., pain and/or itch). For the purposes of in- and exclusion, studies are considered to have induced a placebo or nocebo effect if the (supposed) administration of an inert treatment, is paired with a given learning process attempt to induce positive or negative outcome-effects

Participants/population:

Healthy, adult human volunteers. Patient samples will not be included to improve homogeneity of the results.

Data extraction:

Titles and abstracts of articles retrieved using the search strategy and those from additional sources will be screened by two independent reviewers to identify studies that potentially meet the inclusion criteria outlined above. The full text of these articles and articles about which doubts exist based on the title and/or abstract will be retrieved and assessed for eligibility by two independent reviewers. Full texts that are considered to be possibly eligible for inclusion or about which doubts exist will also be assessed for eligibility by a third reviewer. Two independent reviewers will use a standardized form to extract data from the included studies to derive study characteristics, assess study quality, and for data analysis. Extracted information will include details of the intervention, control condition, study population, sensation type and how sensations were measured (e.g. self-report), type of experimental induction (i.e., learning method used), type of expectancy (i.e., placebo or nocebo), information for quality assessment, and outcome data for meta-analysis (e.g., sample size, mean, and standard deviation). Doubts regarding data-extraction will be resolved through discussion with a second review author. Missing data will be requested from the study authors.

Risk of bias assessment:

Risk of bias will be assessed using the method developed by Marcuzzi and colleagues in 2013 specifically for quantitative sensory testing studies. This method assesses 1) whether the sample was clearly described, 2) whether the sample is representative of the population, 3) whether the somatosensory assessment methods are standardized, validated, and well described, 4) adequate blinding if relevant, and 5) whether potential confounders were taken into account.

Strategy for data synthesis:

A quantitative synthesis, using aggregate data, of the data is planned. The (standardized) mean difference (with a 95% confidence interval) will be calculated for all included studies for which sufficient data are available. Both between and within subject designs will be included; sensitivity analyses will be conducted to test for a difference in design type (within/between). If significant differences are detected, design type will be included in the analyses as a moderator variable). Subsequently, the pooled effects for each of the experimental induction will be analyzed using a random-effects model. The effects of experimental inductions will also be compared between placebo and nocebo effects. If sufficient data are available, the effects of the experimental inductions will be compared between different somatosensory sensations (see below). Where statistical pooling is not possible, the findings of the systematic review will be presented in narrative form. Heterogeneity will be assessed with the I2 statistic, by visual inspection of the forest plot(s), and by subset analyses (see below). The presence of publication bias will also be assessed (e.g., via inspection of a funnel plot).

ELIGIBILITY:
Inclusion Criteria:

* Studies using experimental induction of placebo and/or nocebo effects on somatosensory sensations (i.e., pain and/or itch), which necessitates the (supposed) administration of an inert treatment, which, through a given learning process, is believed to have positive or negative effects.
* This review will include original, controlled experimental studies on healthy participants that employed learning-based inductions of placebo and/or nocebo effects on somatosensory sensations. The studies should be written in English, German or Dutch, available full-text, and published in a peer-reviewed journal. No year restrictions on publication date will be imposed.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Healthy, adult human volunteers. Patient samples will not be included to improve homogeneity of the results.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Placebo magnitude | Through study completion, an average of 1 month
  The magnitude of induced placebo effects, by measures including, but not limited to, self-report measures of perceived sensation intensity or unpleasantness (e.g., as rated on a visual analogue scale or numerical rating scale).
Nocebo magnitude | Through study completion, an average of 1 month
  The magnitude of induced nocebo effects, by measures including, but not limited to, self-report measures of perceived sensation intensity or unpleasantness (e.g., as rated on a visual analogue scale or numerical rating scale).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea WM Evers, Prof. Dr., Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
No personal data are collected, stored, or shared. Data collection is monitored by the department's Data Monitor.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately after publication of the study. Data will be retained for 15 years.
Access Criteria: Data can be shared with scientists in relevant fields for the purpose of future studies such as replication or meta-analysis (or with designated persons for monitoring purposes).

REFERENCES:
- [Derived] Thomaidou MA, Blythe JS, Peerdeman KJ, van Laarhoven AIM, Van Schothorst MME, Veldhuijzen DS, Evers AWM. Learned Nocebo Effects on Cutaneous Sensations of Pain and Itch: A Systematic Review and Meta-analysis of Experimental Behavioral Studies on Healthy Humans. Psychosom Med. 2023 May 1;85(4):308-321. doi: 10.1097/PSY.0000000000001194. Epub 2023 Mar 23. PMID 36961347
- [Derived] Blythe JS, Thomaidou MA, Peerdeman KJ, van Laarhoven AIM, van Schothorst MME, Veldhuijzen DS, Evers AWM. Placebo effects on cutaneous pain and itch: a systematic review and meta-analysis of experimental results and methodology. Pain. 2023 Jun 1;164(6):1181-1199. doi: 10.1097/j.pain.0000000000002820. Epub 2022 Nov 16. PMID 36718994